CLINICAL TRIAL: NCT01852929
Title: The Effect of Sleep Apnea on Sleep Dependent Learning Using the Visual Discrimination Task.
Brief Title: Sleep Apnea and Visual Perceptual Skill Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidi Roth, MD (Other)
Responsible Party: Sponsor-Investigator, Heidi Roth, MD, Associate Professor of Neurology, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 09-1944
Record Dates: First submitted 2013-04-25; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Apnea
Keywords: Memory
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apnea patients on and off PAP in order A (Other): Subject using usual positive airway pressure therapy while sleeping for one night, then crossing over to not using usual apnea therapy while sleeping for another night.
  Interventions: Other: Subject using usual positive airway pressure therapy while sleeping for one night
- Apnea patients on and off PAP in order B (Other): Subject not using apnea therapy while sleeping for one night, then crossing over and subject using usual positive airway pressure therapy while sleeping for one night.
  Interventions: Other: Subject using usual positive airway pressure therapy while sleeping for one night

INTERVENTIONS:
Other: Subject using usual positive airway pressure therapy while sleeping for one night — Participants use their usual positive airway pressure therapy while sleeping overnight

SUMMARY:
The purpose of this study is to determine whether obstructive sleep apnea affects sleep dependent memory and learning. Subjects with apnea will be given a test of perceptual skill learning (the Visual Discrimination Task (VDT)) that has previously been shown to depend on sleep. Subjects will be tested on this task before and after sleep. The difference in performance after sleep compared to before sleep provides a measure of sleep dependent learning. Participants will be tested on one night when they have less apnea because they are using continuous positive airway pressure (CPAP) as prescribed by their physician, which is well known to reduce apnea; and on another night when they are in their native state and have a greater degree of apnea. Memory performance will be compared between the two nights to determine how apnea affects sleep dependent memory.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sleep apnea
* Use PAP therapy as prescribed by his/her physician for 3-4 weeks prior to enrollment
* Right-handed

Exclusion Criteria:

* Major neurological or psychiatric condition
* Chronic pain condition
* Learning disabilities
* Serious brain or head injury (e.g. seizure, stroke, head trauma)
* Major surgery or general anesthesia in the past year
* Pregnant or nursing
* Problems with eyes or vision (besides corrected-to-normal with glasses or contacts)
* Past diagnosis of infection that can affect the brain (e.g. meningitis, HIV/AIDS)
* Medications that affect sleep (antidepressants, muscle relaxants, sleep aids, beta-blockers, stimulants, or corticosteroids)
* Recreational drug use, including marijuana
* Night-shift work
* Cancer or cancer treatment in the last 2 years
* Smoke more than 10 cigarettes per day
* Consume more than 3 caffeinated foods or beverages per day

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
VDT learning Change Score | Change from baseline after 6-9 hours sleep
  Learning on the visual discrimination task (VDT) is measured by comparing performance on the perceptual task at a baseline session prior to sleep to that in a second session after sleep. Subjects are standardly tested in the hour prior to their typical bedtime, and re-tested after spontaneously awakening after a night of sleep. Sleep is known to consolidate learning on this task, such that more robust learning occurs after an interval of sleep compared to when the patient is awake over the same interval (Stickgold et al, J Cog Neurosci,2000; Stickgold et al., Nat Neurosci, 2000). Our aim is to determine if sleep dependent learning is disrupted by apnea, and preserved when apnea is eliminated.

SECONDARY OUTCOMES:
Apnea Hypopnea Index (AHI) | During minimum 6 hour sleep recording
  The AHI is a measure of the average number of respiratory events recorded per hour of sleep based on a record which includes a minimum of 6-hours of recorded sleep. Standard clinical categories for the severity of apnea are as follows: Mild = 5-10/ hour; Moderate = 10-15/ hour; Severe = >15/ hour. We will measure the Apnea Hypopnea Index on the night when participants are using their standard recommended PAP therapy and on the night when they are not using that therapy in order to be able to determine how the degree of apnea (AHI) correlates with the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Roth, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals Sleep Disorders Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Stickgold R, Whidbee D, Schirmer B, Patel V, Hobson JA. Visual discrimination task improvement: A multi-step process occurring during sleep. J Cogn Neurosci. 2000 Mar;12(2):246-54. doi: 10.1162/089892900562075. PMID 10771409
- [Background] Karni A, Sagi D. Where practice makes perfect in texture discrimination: evidence for primary visual cortex plasticity. Proc Natl Acad Sci U S A. 1991 Jun 1;88(11):4966-70. doi: 10.1073/pnas.88.11.4966. PMID 2052578
- [Background] Karni A, Tanne D, Rubenstein BS, Askenasy JJ, Sagi D. Dependence on REM sleep of overnight improvement of a perceptual skill. Science. 1994 Jul 29;265(5172):679-82. doi: 10.1126/science.8036518.
- [Background] Stickgold R, James L, Hobson JA. Visual discrimination learning requires sleep after training. Nat Neurosci. 2000 Dec;3(12):1237-8. doi: 10.1038/81756. No abstract available. PMID 11100141